CLINICAL TRIAL: NCT00104442
Title: Study of the Effects of Current Drug Treatments on Levels of Certain Brain Chemicals in Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CENA713BUS25
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; memory loss; dementia; senility; forgetful; geriatric; behavior; mood swings
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders; Dementia; Behavior | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
Alzheimer's disease is a medical illness that damages the brain and causes problems with memory, mood and behavior. A substance called acetylcholine (ACh), which is naturally produced in the body, plays an important role in the normal functioning of the brain. In subjects with Alzheimer's disease, the level of ACh is greatly reduced. Currently, there are three commonly prescribed drugs used for treating the symptoms of Alzheimer's disease by helping to maintain the level of ACh in the brain. This study will evaluate how much each of these drugs changes the levels of certain brain chemicals that are known to, or may play an important role in, Alzheimer's disease and its symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate Alzheimer's disease
* Must be able to swallow capsule/tablet
* Must have a caregiver who is available to attend all study visits

Exclusion Criteria:

* Digestive problems related to peptic ulcer
* Experienced a heart attack or stroke in the last 6 months
* Serious/unstable asthma or severe pulmonary (lung) disease
* On current treatment with a blood thinner

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Changes in specific brain enzyme activity from baseline to week 13

SECONDARY OUTCOMES:
Correlate changes in specific brain enzyme activity at week 13 to cognition and behavior
Changes in levels of protein biomarkers in Alzheimer's disease and neurodegeneration from baseline to week 13
Correlate changes in specific brain enzyme activity after 13 weeks treatment to changes in global functioning at 13 and 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- See also: Click here for information about study sites in your area — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=306